CLINICAL TRIAL: NCT05393830
Title: The Impact of Insufficient Sleep and Insomnia Disorder on Behavioral and Neural Markers of Emotion Regulation
Brief Title: The Effect of Sleep Loss on Emotion Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Janet M Mullington, PhD, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022P000120
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Sleep; Insomnia; Sleep Deprivation
Keywords: Emotion; Sleep Restriction; Insomnia Disorder; Sleep; Emotion Regulation; functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Independent Groups Comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Sleep (No Intervention): Normal Sleep - Healthy participants are permitted normal nights of polysomnography or actigraphy recorded sleep before participating in an emotion regulation task during functional Magnetic Resonance Imaging (fMRI) scanning
- Sleep Restriction (Active Comparator): Healthy Participants are sleep restricted to 4 hours of sleep for 3 consecutive days before participating in an emotion regulation task during functional Magnetic Resonance Imaging (fMRI) scanning
  Interventions: Behavioral: Sleep Restriction
- Patients with Insomnia Disorder (No Intervention): Patients with Insomnia Disorder will also be recruited and will be permitted normal nights of polysomnography or actigraphy recorded sleep before participating in an emotion regulation task during functional Magnetic Resonance Imaging (fMRI) scanning

INTERVENTIONS:
Behavioral: Sleep Restriction — Three nights of sleep restricted to 4 hours per night.
  Arms: Sleep Restriction

SUMMARY:
The study is designed to investigate the impact of three nights of sleep restricted to 4 hours per night, on the processing and regulation of emotional information compared to Insomnia Disorder and control. The investigators will address and attempt to answer two questions.

(i) How do three nights of reduced sleep or a diagnosis of Insomnia Disorder affect the processing and regulation of emotional information compared to typical, undisturbed sleep? (ii) What overlapping and distinct neural mechanisms are engaged and associated with behavioral effects when attempting to process and regulate emotions in a sleep restricted state or with a clinical diagnosis of Insomnia Disorder? This study will investigate sleep's role in emotion processing and regulation. The findings will help further understanding of the role of sleep in healthy emotional functioning.

DETAILED DESCRIPTION:
Goal 1: How does sleep loss and clinical sleep disruption (i.e. Insomnia Disorder) impact emotion perception and emotion regulation? The investigators are interested in how chronic loss of sleep, either through artificially restricting sleep or clinically related sleep disturbance, impairs our ability to properly perceive and regulate our responses to emotional information using various emotion regulation strategies. There has been research on the effect of sleep loss on broad areas of cognition, such as attention, working memory, and reasoning ability, but the impact of long-term sleep loss on emotional processing and regulation remains largely unexplored. The investigators aim to characterize how sleep loss via experimentally reduced sleep in healthy control participants or clinical sleep disturbance in patients with Insomnia Disorder, affects the ability to accurately perceive emotion. Investigators will also investigate how it alters the intensity with which emotions are perceived, and the effect that these changes have on the ability to regulate emotional responses to these stimuli compared to healthy control participants that are allowed undisturbed sleep.

Goal 2: How are changes in subjective emotional responses reflected in the neural signal and psychophysiological measures? The investigators will utilize fMRI and measures of autonomic reactivity (heart rate and skin conductance) to characterize the neural and psychophysiological responses that are associated with behavioral changes following sleep restriction or in patients with Insomnia disorder compared to healthy sleep control participants.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to follow the protocol
* willing and able to meet inclusion criteria for fMRI scanning
* willing to refrain from alcohol and recreational drugs for the duration of the protocol
* normal or corrected to normal vision is required

Exclusion Criteria:

* left-handedness or ambidexterity
* the use of any drugs that could affect either sleep or cognitive functioning (e.g., prescription sleeping pills or antidepressants)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Emotional Regulation Task with Strategy | Day 1
  Baseline behavioral ratings to emotional stimuli with emotion regulation strategies
Baseline Emotional Regulation Task without Strategy | Day 1
  Baseline behavioral ratings to emotional stimuli without emotion regulation strategies
Reassessment of the Emotional Regulation Task with Strategy Baseline behavioral ratings to emotional stimuli with or without emotion regulation strategies | one test in a 3-6 day window
  Behavioral ratings to emotional stimuli with emotion regulation strategies following normal sleep or sleep restriction
Reassessment of the Emotional Regulation Task without Strategy Baseline behavioral ratings to emotional stimuli with or without emotion regulation strategies | one test in a 3-6 day window
  Behavioral ratings to emotional stimuli without emotion regulation strategies following normal sleep or sleep restriction

SECONDARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | one test in a 3-6 day window
  fMRI measured neural reactivity (blood oxygen-level dependent signal)

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Mullington, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We are developing our institutional data sharing plan